CLINICAL TRIAL: NCT05568017
Title: Neoadjuvant Peptide Receptor Radionuclide Therapy (PRRT) With 90Y-DOTATOC in Pancreatic Neuroendocrine Tumours.
Brief Title: Neoadjuvant PRRT With Y-90-DOTATOC in pNET
Acronym: NeoNet
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty in recruiting patients also due to the pandemic period, presence of competitive studies.
Sponsor: European Institute of Oncology (Other)
Collaborators: Agenzia Italiana del Farmaco (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IEO 906
Record Dates: First submitted 2022-09-23; First posted 2022-10-05 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2022-09

CONDITIONS: Pancreatic Neuroendocrine Tumor
MeSH Terms: conditions — Adenoma, Islet Cell

STUDY DESIGN:
Intervention Model Description: Patients affected by unresectable or borderline resectable P-NETs and limited liver disease will be enrolled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Y-90-DOTATOC (Experimental): Patients will receive PRRT with Y-90-DOTATOC
  Interventions: Drug: peptide receptor radionuclide therapy with Y-90-DOTATOC

INTERVENTIONS:
Drug: peptide receptor radionuclide therapy with Y-90-DOTATOC — Patients with unresectable or borderline resectable pNETs will recive PRRT with 90Y-DOTATOC
  Other Names: PRRT; Y-90-DOTATOC

SUMMARY:
Neuroendocrine tumors (NETs) are relatively rare tumors, mainly originating from the digestive system, that tend to be slow growing and are often diagnosed when metastatic. Surgery is the sole curative option, but is feasible only in a minority of patients.

Peptide Receptor Radionuclide Therapy (PRRT) has been experimented for almost 20 years and is an established effective therapeutic modality for well/moderately differentiated, inoperable or metastasized gastro-entero-pancreatic (GEP) and bronchial NETs. Clinical studies demonstrated that partial and complete objective responses can be obtained in up to 30% of patients. Side effects may involve the kidneys and the bone marrow and are usually mild. Renal protection is used to minimize the risk of a late decrease of renal function.

A new application for P-NETs is preoperative PRRT. Since surgery is the only curative option for GEPNETs, preoperative PRRT could increase the efficacy of surgery. However, this modality has not been fully explored in dedicated studies and there are just few sporadic case reports that described the preoperative use of PRRT in pancreatic NETs who could then be operated on successfully. Moreover there are few experiences demonstrating the advantage of PRRT associated to surgery in a multidisciplinary setting. In addition, the possibility of detecting the circulating NET transcripts by means of transcriptome analysis could represent an early marker of response to PRRT and improve the patient management.

Aim of this study is to evaluate the response and rate of R0 surgery in patients with unresectable or borderline resectable PNETs eligible to PRRT with 90Y-DOTATOC and correlate the response to the variation in circulating NET transcripts measured before and after the end of PRRT. It has been recently shown that a PCR-based 51 transcript signature is significantly more sensitive and efficient than single analytes (e.g. CgA) in NET diagnosis and follow up.

30 patients will be enrolled in the study; each of them will receive 1.85 GBq/cycle of 90Y-DOTATOC with a cumulative activity of 9.25-11.1 GBq in 5-6 cycles (depending on personalized dosimetry). Therapy response will be assessed by morphological (CT/MRI) and functional (PET/CT or Octreoscan) imaging after 3 and 6 months from the completion of PRRT and compared with transcript analysis.

Based on literature reports we expect a response rate of about 35% of patients.

DETAILED DESCRIPTION:
GEP-NETs tend to be slow growing (although aggressive forms exist) and are often diagnosed when they have already metastasized, when a radical treatment is no longer possible.

Treatment of NETs is typically multidisciplinary and should be individualized according to tumor type, burden, and symptoms. Therapeutic tools include surgery, interventional radiology and medical treatments such as somatostatin analogues, interferon, chemotherapy, new targeted drugs and peptide receptor radionuclide therapy (PRRT) with radiolabeled somatostatin analogues [Modlin 2008]. Several clinical trials have indicated that PRRT with somatostatin analogues 90Y-DOTATOC, 177Lu-DOTATATE and 177Lu-DOTATOC, is an efficient tool in the management of NETs (30% objective responses with a great survival benefit) which compares favorably to classic chemotherapy results (up to 20% responses) [Kwekkeboom 2005].

Dosimetric studies demonstrated that these radiopeptides are able to deliver high radiation doses to somatostatin receptor sst2-expressing tumors and acceptable doses to normal organs [Cremonesi 2010]. Side effects, usually mild, may involve kidneys and bone marrow. Renal protection is used to minimize the risk of a late function decrease [Bodei 2003].

Pts are selected for PRRT based on molecular imaging with 111In-pentetreotide or, more recently, a 68Ga-SSA-PET, such as 68Ga-DOTATOC/DOTATATE/DOTANOC [Virgolini 2010], which have revolutionized the NET imaging, with an overall sensitivity of >90%, and specificity ranging from 92% to 98% [Ambrosini 2012].

PRRT is an innovative therapeutic approach for inoperable or metastasized, well/moderately differentiated GEP and bronchial NETs. PRRT in P-NETs has demonstrated efficacy in terms of objective response and impact on survival parameters. Since surgery is the only curative option for patients with GEP-NETs, it is proposed that neoadjuvant treatment will improve outcome by enabling disease regression that will enable surgical resection.

Identification of disease regression as assessed by a PCR-blood based analysis of circulating neuroendocrine tumor transcripts will provide objective and quantifiable molecular genomic early information that is additive to imaging criteria of regression. This will objectively establish PRRT treatment efficacy and thereby facilitate the identification and selection of individuals that would then benefit from surgical intervention.

The two most commonly used radiopeptides, 90Y-DOTATOC and 177Lu-DOTATATE, produce overall objective response rates of 15-35%. Particularly relevant is the outcome in terms of both progression-free and overall survivals, which compare favorably with biotherapies. PRRT is generally well tolerated with mild toxicity, if the necessary precautions, such as the co-administration of nephron-protective amino acids or the adjustment of the administered activity, are taken.

PRRT in P-NETs has demonstrated efficacy in terms of objective response and impact on survival parameters. Response rates are >35%, higher than in small intestine tumors. In particular, in 342 patients with P-NETs, out of the whole series of 1109 patients treated with 90Y-DOTATOC, 47% objective responses were reported by Imhof in 2011. In 2013, Sansovini reported 39% partial and complete responses using 177Lu-DOTATATE at full dosage, while 60.3% partial responses were reported by Ezziddin in 2014 using the same peptide. Reported progression free survival (PFS) rates are > 30 months.

An interesting new application for P-NETs is the neoadjuvant setting, which was suggested by sporadic case reports that described the successful surgical resection in patients with initially inoperable P-NETs treated with PRRT. However, this treatment modality has not been fully explored in dedicated studies.

Moreover, there are few experiences demonstrating the advantage of PRRT associated to surgery in a multidisciplinary setting [Bertani 2014, 2016].

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by unresectable or borderline resectable P-NETs and limited liver disease
* Multidisciplinary evaluation in which a global therapy approach is proposed with PRRT in a neoadjuvant setting.
* Histopathologic diagnosis of WHO G1/G2 P-NET
* Conserved hematological, liver and renal parameters: hemoglobin >/= 10 g/dL, absolute neutrophil count (ANC) >/= 1.5 x 109 /L, platelets >/= 100 x 109 /L, bilirubin </= 1.5 X UNL (upper normal limit), ALT < 2.5 X UNL (< 5 X UNL in presence of liver metastases), creatinine < 2 mg/dL.
* Age more than 18 years.
* Patients with documented disease will be admitted to therapeutic phase only if the diagnostic receptor imaging (Ga-68-peptides PET/CT or OctreoScan) demonstrate a significant uptake in the tumor (grade 2 or 3, according to a preset scoring, where grade 1= equal to normal liver, grade2 = higher than normal liver, grade 3= higher than kidneys and spleen), that may allow delivering a low absorbed dose to normal organs and a high dose to the tumor [Cremonesi 1999, Cremonesi 2010].
* Disease must be measurable by means of conventional imaging (CT or MRI)
* Before treatment clinical history data will be collected, physical examination will be performed and diagnostic and laboratory data will be examined.
* Patients must not receive other treatments (e.g. chemo- or radiotherapy) from one month before to two months after the completion of 90Y-DOTATOC cycles.
* Patients must be naive from previous radionuclide treatments with radiopeptides (e.g. 111Inpentetreotide, Lu-177-petides) or other radiopharmaceuticals (e.s. 131I-MIBG, 131I).

Exclusion Criteria:

* - Pregnancy/breastfeeding (a pregnancy test not older than 7 days is mandatory).
* Assessed bone marrow invasion > 25%.
* Other concomitant neoplasm (excluding in situ basaliomas and radically treated cervical cancers).
* ECOG score higher than 2.
* Expectancy of life shorter than 6 months.
* Patients with psycho-physical conditions that are not suitable for entering this clinical study and fulfilling its requirements.
* No multidisciplinary indication to surgery after PRRT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2022-09-23 (Actual); Study Completion 2024-11-11 (Actual)

PRIMARY OUTCOMES:
objective response evaluation | 3 months after end of PRRT
  objective responses (partial and complete responses, stable disease) will be evaluated according to modified RECIST criteria (mRECIST).
objective response evaluation | 6 months after end of PRRT
  objective responses (partial and complete responses, stable disease) will be evaluated according to modified RECIST criteria (mRECIST).

SECONDARY OUTCOMES:
rate of operability | 3 months after the end of PRRT.
  to evaluate the rate of operability 3 months after the end of PRRT.
rate of operability | 3 months after the end of PRRT.
  to evaluate the rate of operability 6 months after the end of PRRT.
analysis of tumor specific circulating NET transcripts | before PRRT, and 3 and 6 months after therapy.
  Assess the response to PRRT by means of a neuroendocrine tumor specific PCR-blood based multianalyte molecular algorhythmic analysis of circulating NET transcripts

CONTACTS AND LOCATIONS:
Locations (1):
- Chiara Maria Grana, Milan, Italy

IPD SHARING:
Plan to Share IPD: No